CLINICAL TRIAL: NCT05918458
Title: Pulmonary Hypertension Clinical Trials: What Are Prevailing Patient Experiences in Pulmonary Hypertension Studies
Brief Title: Discovering Clinical Study Experiences of Patients With Pulmonary Hypertension
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82814554
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of pulmonary hypertension patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future pulmonary hypertension patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Able to comprehend the investigational nature of the protocol and provide informed consent
* Diagnosis of pulmonary hypertension

Exclusion Criteria:

* No diagnosis of pulmonary hypertension confirmed
* Inability to perform regular electronic reporting
* Patient does not understand, sign, and return consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary hypertension who are actively considering enrolling in an interventional clinical trial for said condition, but have not yet completed enrollment and randomization phases in said clinical trial.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in a pulmonary hypertension clinical research | 3 months
Rate of patients who remain in pulmonary hypertension clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jais X, Brenot P, Bouvaist H, Jevnikar M, Canuet M, Chabanne C, Chaouat A, Cottin V, De Groote P, Favrolt N, Horeau-Langlard D, Magro P, Savale L, Prevot G, Renard S, Sitbon O, Parent F, Tresorier R, Tromeur C, Piedvache C, Grimaldi L, Fadel E, Montani D, Humbert M, Simonneau G. Balloon pulmonary angioplasty versus riociguat for the treatment of inoperable chronic thromboembolic pulmonary hypertension (RACE): a multicentre, phase 3, open-label, randomised controlled trial and ancillary follow-up study. Lancet Respir Med. 2022 Oct;10(10):961-971. doi: 10.1016/S2213-2600(22)00214-4. Epub 2022 Aug 1. PMID 35926542
- [Background] Divers C, Platt D, Wang E, Lin J, Lingohr-Smith M, Mathai SC. A Review of Clinical Trial Endpoints of Patients with Pulmonary Arterial Hypertension and Chronic Thromboembolic Pulmonary Hypertension and How They Relate to Patient Outcomes in the United States. J Manag Care Spec Pharm. 2017 Jan;23(1):92-104. doi: 10.18553/jmcp.2017.23.1.92. PMID 28025931
- [Background] Harder EM, Waxman AB. Clinical trials in group 3 pulmonary hypertension. Curr Opin Pulm Med. 2020 Sep;26(5):391-396. doi: 10.1097/MCP.0000000000000694. PMID 32657833

DOCUMENTS (1):
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05918458/ICF_000.pdf